CLINICAL TRIAL: NCT04251884
Title: Pudendal Nerve Block in Patient Treated for Hemorrhoidectomy Under Spinal Anaesthesia: Prospective Randomized Double-blind Controlled Trial
Brief Title: Pudendal Nerve Block for Hemorrhoidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Francesco Mongelli (Other)
Responsible Party: Sponsor-Investigator, Francesco Mongelli, MD, Ospedale Regionale Bellinzona e Valli
Organization: Ospedale Regionale Bellinzona e Valli (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE TI 3222
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Results first posted 2020-06-05 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Hemorrhoids; Postoperative Pain
MeSH Terms: conditions — Hemorrhoids; Pain, Postoperative | interventions — Anesthetics, Local; Ropivacaine

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Receiving the pudendal nerve block (Experimental)
  Interventions: Procedure: Local anesthetic (ropivacaine)
- Not receiving the pudendal nerve block (Active Comparator)
  Interventions: Procedure: Local anesthetic (ropivacaine)

INTERVENTIONS:
Procedure: Local anesthetic (ropivacaine) — Patients randomized in the treatment arm will receive a sonography-guided pudendal nerve block
  Other Names: No pudendal nerve block

SUMMARY:
Patients undergoing Milligan-Morgan hemorrhoidectomy will be randomized to receive or not the pudendal nerve block after the spinal anesthesia.

DETAILED DESCRIPTION:
Patients included were those undergoing Milligan-Morgan hemorrhoidectomy under spinal anaesthesia from January 2018 to December 2019. Exclusion criteria were age < 18 years old, pregnancy and allergy to local anaesthetics. Patients meeting inclusion and exclusion criteria were randomized to undergo an ultrasound-guided pudendal nerve block. Per-protocol all patients received postoperative metronidazole 500 mg for 3 days, laxative, a basis analgesia with NSAID and opioids as needed. Postoperative pain on the visual analogue scale (VAS) at 6, 12, 24 and 48 hours, opioids needed, complications and length of hospital stay were recorded. Patients and ward personnel were not informed about the treatment arm. All Patients were further controlled 6 weeks after the intervention.

ELIGIBILITY:
Inclusion criteria:

* Patients affected by haemorrhoids (grade III and IV) and treated with Milligan-Morgan hemorrhoidectomy under spinal anaesthesia
* Signed informed consent

Exclusion criteria:

* Age < 18 years old
* Pregnancy
* Allergy to local anaesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-29 (Actual); Study Completion 2020-01-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Regionale di Bellinzona e Valli, Bellinzona, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Di Giuseppe M, Saporito A, La Regina D, Tasciotti E, Ghielmini E, Vannelli A, Pini R, Mongelli F. Ultrasound-guided pudendal nerve block in patients undergoing open hemorrhoidectomy: a double-blind randomized controlled trial. Int J Colorectal Dis. 2020 Sep;35(9):1741-1747. doi: 10.1007/s00384-020-03630-x. Epub 2020 May 30. PMID 32474710

RESULTS

PARTICIPANT FLOW:
Groups:
- Receiving the Pudendal Nerve Block: Ultrasound-guided pudendal nerve block performed with 20 mls Ropivacaine 0.75%.
- Not Receiving the Pudendal Nerve Block: No ultrasound-guided pudendal block performed
Period: Overall Study
Arm/Group | Receiving the Pudendal Nerve Block | Not Receiving the Pudendal Nerve Block
Started | 23 | 26
Completed | 23 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Not Receiving the Pudendal Nerve Block: No ultrasound-guided pudendal nerve block performed.
- Total: Total of all reporting groups
Arm/Group | Receiving the Pudendal Nerve Block | Not Receiving the Pudendal Nerve Block | Total
Number analyzed (Participants) | 23 | 26 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (18.3) | 53.3 (17.5) | 52.5 (17.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 12 | 15 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Switzerland | 23 | 26 | 49
Comorbidities (Cardiologic, Pulmonary, Kidney, Diabetes, Neuropathy) [Number; unit: participants]
  • Cardiologic disease | 2 | 3 | 5
  • Pulmonary disease | 0 | 3 | 3
  • Kidney disease | 2 | 1 | 3
  • Diabetes | 1 | 2 | 3
  • Neuropathy | 0 | 1 | 1
Symptoms leading to surgery (itching, pain, bleeding, tenesmus) [Number; unit: participants]
  Itching | 10 | 9 | 19
  Pain | 20 | 23 | 43
  Bleeding | 12 | 19 | 31
  Tenesmus | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain on the Visual Analogue Scale (VAS)
Description: Visual analogue scale (VAS) ranges from 0 to 10, where 0 is "no pain at all" and 10 is "the strongest pain"
Time Frame: at 24 hours after the hemorrhoidectomy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Receiving the Pudendal Nerve Block | Not Receiving the Pudendal Nerve Block
Number analyzed (Participants) | 23 | 26
units on a scale | 1.4 (1.4) | 3.1 (2.4)

2. Secondary Outcome: Postoperative Pain on the Visual Analogue Scale (VAS)
Description: Visual analogue scale (VAS) ranges from 0 to 10, where 0 is "no pain at all" and 10 is "the strongest pain"
Time Frame: at 6, 12 and 48 hours after the operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Receiving the Pudendal Nerve Block | Not Receiving the Pudendal Nerve Block
Number analyzed (Participants) | 23 | 26
score on a scale
  Pain on VAS at 6 hours | 2.8 (2.4) | 4.6 (3.7)
  Pain on VAS at 12 hours | 3.4 (3.1) | 4.7 (3.6)
  Pain on VAS at 48 hours | 1.0 (1.6) | 2.1 (2.0)

3. Secondary Outcome: Opioids Consumption
Time Frame: Within 48 hours
Measure: Count of Participants; unit: Participants
Groups:
- Receiving the Pudendal Nerve Block: Ultrasound-guided pudendal nerve block with performed 20 mls Ropivacaine 0.75%.
Arm/Group | Receiving the Pudendal Nerve Block | Not Receiving the Pudendal Nerve Block
Number analyzed (Participants) | 23 | 26
Participants | 5 | 10

4. Secondary Outcome: Lenght of Hospital Stay
Time Frame: up to 2 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Receiving the Pudendal Nerve Block | Not Receiving the Pudendal Nerve Block
Number analyzed (Participants) | 23 | 26
days | 1.2 (1.2) | 1.8 (1.8)

5. Secondary Outcome: Complications Related to the Pudendal Nerve Block
Time Frame: Within 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Receiving the Pudendal Nerve Block | Not Receiving the Pudendal Nerve Block
Number analyzed (Participants) | 23 | 26
Participants | 0 | 0

6. Secondary Outcome: Direct and Indirect Cost Analysis in Out- and In-patients
Description: Ongoing
Time Frame: Within the hospital stay
Reporting Status: Not Posted, anticipated posting 2022-09

ADVERSE EVENTS:
Time Frame: 2 years
Description: Any adverse event related to the pudendal nerve block.
Arm/Group | Receiving the Pudendal Nerve Block | Not Receiving the Pudendal Nerve Block
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/26
Other Adverse Events (participants affected / at risk) | 0/23 | 0/26

LIMITATIONS AND CAVEATS:
The main limitation of the study was represented by the small number of enrolled patients and larger sample are required to confirm our results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/84/NCT04251884/Prot_SAP_000.pdf